CLINICAL TRIAL: NCT04225208
Title: A Phase I, Single-centre, Non-Randomised, Open-label, Pharmacokinetic and Mass Balance Study of Orally Administered [14C]-AZD4205 in Healthy Adult Male Subjects
Brief Title: Pharmacokinetic and Mass Balance Study of Orally Administered [14C]-AZD4205 in Healthy Adult Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dizal Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DZ2019J0002
Record Dates: First submitted 2020-01-03; First posted 2020-01-13 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2019-12

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Single Person

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [14C]-AZD4205 (Experimental): A single dose of [14C]-AZD4205
  Interventions: Drug: [14C]-AZD4205, single 50 mg oral dose administrated on day 1

INTERVENTIONS:
Drug: [14C]-AZD4205, single 50 mg oral dose administrated on day 1 — Each subject will receive 50 mg AZD4205 oral solution (free base equivalent) containing a nominal dose of 15 µCi [14C]- radiolabelled AZD4205 as a single administration .

SUMMARY:
This is a phase I, open label, healthy volunteers, ADME study with single oral administration of [14C]-AZD4205.

DETAILED DESCRIPTION:
Phase I study to evaluate the excretion of AZD4205 radioactive dose, the metabolic profile, pharmacokinetics, safety and tolerability following a single oral administration of [14C]-AZD4205 in healthy male volunteers. The purpose of this study is to investigate ADME properties of AZD4205 by analyzing blood, urine and feces collected during the study

ELIGIBILITY:
Inclusion Criteria:

* 1. Healthy male subjects aged 18 to 65, who must be willing to use reliable methods of contraception, even if their partners are postmenopausal, surgically sterile, or using an effective hormonal method of contraception or intrauterine coil.
* 2. In addition, subjects must agree to continue to take similar contraceptive precautions until 6 months after administration of AZD4205 and avoid procreative sex as well as sperm donation for 6 months after administration of AZD4205.

Exclusion Criteria:

* 1. Any clinically relevant abnormalities in physical examination, vital signs, hematology, clinical chemistry, urinalysis or ECG at screening or baseline in the opinion of the investigator.
* 2. Subjects who may have been exposed to radiation for therapeutic or diagnostic reasons at levels above background (e.g,, through X-ray examination other than dental X-rays or plain X-rays of thorax or bony skeleton) of > 5 mSv in last year, > 10 mSv over last 5 years or a cumulative total of > 1 mSv per year of life.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 8 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2020-03-02 (Actual)

PRIMARY OUTCOMES:
Percentage of radioactive dose recovered in urine and faeces and total percentage | Up to 57 days
  To evaluate the percentage of radioactive dose of [14C] radiolabelled AZD4205 recovered in urine, feces, and in total
Provide samples for subsequent studies | Up to 57 days
  Provide samples for subsequent studies to characterize the metabolism of [14C]AZD4205

SECONDARY OUTCOMES:
AUC(0-inf) for [14C] radioactivity in plasma and whole blood | Up to 57 days
  To determine AZD4205 plasma concentrations and the resulting AUC(0-inf)
AUC(0-t) for [14C] radioactivity in plasma and whole blood | Up to 57 days
  To determine AZD4205 plasma concentrations and the resulting AUC(0-t)
Cmax for [14C] radioactivity in plasma and whole blood | Up to 57 days
  To determine AZD4205 plasma concentrations and the resulting Cmax
tmax for [14C] radioactivity in plasma and whole blood | Up to 57 days
  To determine AZD4205 plasma concentrations and the resulting tmax
tlag for [14C] radioactivity in plasma and whole blood | Up to 57 days
  To determine AZD4205 plasma concentrations and the resulting tlag
t1/2 for [14C] radioactivity in plasma and whole blood | Up to 57 days
  To determine AZD4205 plasma concentrations and the resulting t1/2
λz for [14C] radioactivity in plasma and whole blood | Up to 57 days
  To determine AZD4205 plasma concentrations and the resulting λz
CL/F for [14C] radioactivity in plasma and whole blood | Up to 57 days
  To determine AZD4205 plasma concentrations and the resulting CL/F
Vss/F for [14C] radioactivity in plasma and whole blood | Up to 57 days
  To determine AZD4205 plasma concentrations and the resulting Vss/F
Distribution of total radioactivity in blood | Up to 57 days
  To compare disposition of drug-related total radioactivity in whole blood to that in plasma

OTHER OUTCOMES:
Number of participants with treatment-related adverse events, and serious adverse events | Up to 57 days
  To assess the safety and tolerability of a single dose of AZD4205 in healthy adult male subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Royce Morrison, Principal Investigator — Pharmaron CPC
Locations (1):
- Pharmaron CPC, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No